CLINICAL TRIAL: NCT06468670
Title: Short-course Radiotherapy Combined With Sintilimab for Neoadjuvant Treatment of Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeoES-ljc
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- short-course radiotherapy+sintilimab (Experimental)
  Interventions: Drug: sintilimab，programmed death 1 monoclonal antibody

INTERVENTIONS:
Drug: sintilimab，programmed death 1 monoclonal antibody — short-course radiotherapy
  +sintilimab (200mg, iv, D1, Q3W)

SUMMARY:
This study is aimed to evaluate the efficacy and safety of short-course radiotherapy combined with sintilimab in neoadjuvant treatment of stage III, locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study was designed as a single arm, phase II trial. Subjects will receive short-course radiotherapy combined with sintilimab as neoadjuvant therapy of stage III, locally advanced esophageal squamous cell carcinoma. The primary endpoint is pathologic complete response(pCR).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and ≤75 years old

  * Esophageal squamous cell carcinoma diagnosed biopsy histopathology
  * Patients with resectable esophageal squamous cell carcinoma confirmed by pathology (including histology or cytology) , with pathological stage T3-4 or N+
  * At least one measurable lesion
  * Eastern cooperative oncology group (ECOG) performance status of 0 to 1
  * With adequate organs function

Exclusion Criteria:

* Patients with active malignancy within 5 years other than the tumor studied in this study or a localized tumor that has been cured such as resected basal or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or breast cancer
* Patients who have a higher risk of bleeding or perforation due to the tumor's obvious invasion of the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed a fistula
* Patients who have received any anti-tumor therapy for the research disease in the past, including radiotherapy, chemotherapy, immunotherapy (including but not limited to interleukin, interferon, thymus hormone) and traditional Chinese medicine therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 4 weeks after surgery
  Total tumor regression rate under pathologyPrimary tumor or lymph node surgery specimen pathological examination without residual tumor cell
Incidence rate of adverse events | 3 years
  The ratio of the number of cases with adverse events to the total number of cases available for evaluation.

SECONDARY OUTCOMES:
overall survival | 3 years
  the time from randomization to death
Disease-free survival | 3 years
  the time from treatment until the recurrence of disease (or death) after undergoing curative-intent treatment

IPD SHARING:
Plan to Share IPD: No